CLINICAL TRIAL: NCT01951079
Title: The Safety and Outcome of Intra-amniotic DIGOXIN Injection for Feticide Prior to Second Trimester Abortion
Brief Title: Intra Amniotic Injection of DIGOXIN for Feticide in Second Trimester Termination of Pregnancy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC130077-12CTIL
Record Dates: First submitted 2013-07-16; First posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Arrhythmia; ECG Changes; Hypotension
Keywords: Digoxin; Intra-amniotic injection; feticide; second trimester abortion
MeSH Terms: conditions — Arrhythmias, Cardiac; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- second trimester abortion , feticide (Experimental): all patients admitting to second trimester abortion above 22 weeks will be injected intra-amniotic DIGOXIN for feticide .
  Interventions: Drug: Intra-amniotic injection of DIGOXIN

INTERVENTIONS:
Drug: Intra-amniotic injection of DIGOXIN

SUMMARY:
In second trimester abortion above 22 weeks the investigators usually inject intra-cardiac Kcl for feticide. Digoxin intra-amniotic injection has been described in the literature in doses of 1-1.5 mg. with a success rate of about 80%, and up to 24 weeks. Our aim in this study is to investigate the safety and success rate of 1.5-2 mg. digoxin, intra-amniotic up to 30 weeks pregnancy .

DETAILED DESCRIPTION:
* The digoxin will be injected intra-amniotic with U.S guided, trying to avoid any placental passage or intravascular injection /
* Any patient will have prior to the procedure a full examination including E.C.G and cardiac clearance.

ELIGIBILITY:
Inclusion Criteria:

* healthy women with no medical, cardiac, hypertension, liver or renal problems - pregnant in their 20-30 week gestation,
* that need to have abortion due to fetal anomalies or any other reason
* need to have feticide prior to the procedure

Exclusion Criteria:

* any patient with medical problem that may be a contra-indication to Digoxin
* cardiac problems,
* prior cardiac surgery,
* liver or kidney disease,
* hyper tension etc.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Efficiency of intra-amniotic Digoxin injection for second trimester feticide | a year
  To measure the Success rate of intra-amniotic Digoxin injection for feticide prior to second trimester abortion

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Dr. Zvi Klein, Kfar Saba
  - Sapir medical center, Kfar Saba